CLINICAL TRIAL: NCT03851380
Title: Targeting Functional Improvement in rTMS Therapy
Brief Title: Improving Brain Stimulation Through Imaging
Acronym: IBSI
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Providence VA Medical Center (U.S. Federal Agency); Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D3152-R; 48212 (Other: Stanford IRB)
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Depression; Depressive Disorder, Treatment-Resistant; COVID Stress
Keywords: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Functional Magnetic Resonance Imaging; fMRI; TMS; Neuronavigation; MRI; Transcranial Electrical Stimulation; COVID Stress
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Treatment Resistant Major Depression: Patients with treatment resistant major depression
  Interventions: Behavioral: Psychological / Functional Assessment; Other: Structural and Functional MRI; Device: Transcranial Magnetic Brain Stimulation and MR Image Guidance
- COVID Stress: Veterans with COVID-19-related distress
  Interventions: Behavioral: Psychological / Functional Assessment; Other: Structural and Functional MRI; Device: Transcranial Electrical Stimulation (tES)

INTERVENTIONS:
Behavioral: Psychological / Functional Assessment — Psychological and functional assessment battery to characterize participants.
Other: Structural and Functional MRI — Structural and functional magnetic resonance imaging session.
Device: Transcranial Magnetic Brain Stimulation and MR Image Guidance — MRI guided transcranial magnetic stimulation and measurement of targeting accuracy.
  Groups: Treatment Resistant Major Depression
Device: Transcranial Electrical Stimulation (tES) — Home-based Transcranial Direct Current Stimulation
  Groups: COVID Stress

SUMMARY:
Repetitive pulse transcranial magnetic stimulation (rTMS) is a noninvasive treatment that involves stimulating the brain; however, treatment benefit depends on placing a TMS coil in the correct place on the head to reach critical brain regions below. Clinicians typically use scalp-based targeting, a process in which rather than using MRI guidance to target brain regions for stimulation, they use landmarks on the scalp. Several researchers, including the investigators' lab, showed that the current scalp-based targeting techniques do not position stimulation above the correct brain region, and patients fail to respond. The investigators propose to improve clinical scalp-based targeting by comparing it to MRI guided targeting. The most common clinical population receiving rTMS therapy is depressed patients. The investigators' plan is to study the accuracy of certain scalp-based rules in patients with depression. Accurate brain stimulation targeting is critical for effective rTMS therapy.

For participants who are not undergoing rTMS therapy who have COVID-19 distress, we are offering a combined home-based neuromodulation (transcranial electrical stimulation) and focused psychotherapy program dedicated to improving the same outcome measure, quality of life. Transcranial electrical stimulation (tES) stimulates the brain over a large region; however, we are able to model with brain imaging which brain regions receive the strongest stimulation. Our goal is still to examine stimulation precision, but we will test whether strength of tES in the same brain regions that rTMS is targeting will also lead to improved quality of life. We will also carefully assess whether it is possible to measure healthy functioning, an outcome in the rTMS study, because sheltering in place may reduce activities and thus distort our measure. We will also test whether our psychotherapy intervention will mitigate this effect and, if so, we may make it available to all those depressed Veterans in whom we're studying the effect of neuromodulation on functioning.

DETAILED DESCRIPTION:
Potential participants are first identified and contact is made. Potential participants are then screened for inclusionary and exclusionary information (see tab 9. Eligibility) that relate to whether they can safely and comfortably perform the procedures and whether they are considered healthy or have the disorder for which brain stimulation therapy will be delivered. They will undergo informed consent that will disclose all the different risks and benefits for the procedures they will undergo. The list of procedures in which participants consent to participate is below. Participants may do either or both of the activities detailed below.

PROCEDURES:

For participants in the MRI guided targeting activity:

1. Psychological / functional assessments:

   Interview, computerized, and paper and pencil measures of psychological functioning. These measures are used to characterize patients' diagnosis and psychological status. For example, depressed patients will answer questions about depressive symptoms and potentially comorbid symptoms such as post-traumatic stress disorder. This testing typically lasts 2 hours.
2. MRI and functional MRI Patients will undergo an MRI that indicates where they receive stimulation by a marker placed on a cap that displays brightly on an MRI. MRI will occur at Lucas center or the Palo Alto VA and involves brain imaging that will be related to brain stimulation techniques either through facilitating image guidance or providing information that will be correlated to data collected during stimulation. Typically, a session lasts about 2.5 hours since there is setup time involved.
3. Brain Stimulation:

TMS-transcranial magnetic stimulation which will be collected at the Palo Alto VA. Part of this procedure may include electromyography (EMG) which involves placing electrodes on the skin, typically the hand, and measuring indicators of muscle contraction. Sometimes this information is used to decide stimulation intensity during TMS and sometimes the TMS induced response will be a source of data in itself. Typically, this is only a measure conducted in parallel with other procedures and thus will not be given its own consent. MRI Guided TMS. An MRI will be used to target a selective brain region. To accomplish this, the MRI will be displayed on a computer screen and an infrared camera enables identification of the correspondence between the image and the participant's head. To study errors in scalp-based targeting, the investigators will perform scalp targeting while under MRI guidance but without the typical visual feedback provided by the MRI. Then this will be compared to scalp targeting with MRI guidance. The difference will identify typical errors in scalp targeting. Typically, a session will last approximately 1.5 hours.

For participants in the home-based neuromodulation and focused psychotherapy program:

1. Psychological / functional assessments:

   Interview, computerized, and paper and pencil measures of psychological functioning. These measures are used to characterize patients' diagnosis and psychological status. For example, depressed patients will answer questions about depressive symptoms and potentially comorbid symptoms such as post-traumatic stress disorder. This testing typically lasts 2 hours.
2. MRI and functional MRI Patients will undergo an MRI that indicates where they receive stimulation by a marker placed on a cap that displays brightly on an MRI. At Lucas center or the Palo Alto VA and involves brain imaging that will be related to brain stimulation techniques either through facilitating image guidance or providing information that will be correlated to data collected during stimulation. Typically, a session lasts about 2.5 hours since there is setup time involved.
3. Transcranial Electrical Stimulation (tES) and Therapy Transcranial electric stimulation (tES) is a brain stimulation technique in which two electrodes will be placed on the participant's scalp and a weak, painless electrical current will be passed between the electrodes. These sessions will occur daily and last about 30 minutes. This protocol also integrates neuromodulation with stress management since combined stimulation and therapy have been demonstrated to be more effective. During tES, participants will practice meditation/relaxation/self-quieting using biofeedback (e.g. hand temperature monitoring). Participants will also receive weekly stress-management skills training. For participants with COVID-19 related stress, we will include specialized examples from a COVID-19 specialized therapy. During the meditation/relaxation/self-quieting, the participant will be asked to listen to a scripted recording or, in the event they do not like the recording or do not find it relaxing, they may negotiate an alternative with the study team (e.g. 30 minutes of classical music).
4. Actigraphy Participants undergoing tES would be required to wear a watch-like device for 6 weeks during tES therapy that functions much like a "Fitbit" to measure their sleep and activity.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

Capacity and willingness to participant in TMS, and fMRI as well as satisfying criteria for diagnosis.

* Between 18 and 89 years of age.
* Ability to obtain a Motor Threshold (MT) with single pulse TMS
* Ability to safely and comfortably undergo an MRI and TMS
* Able to read, verbalize, understand and voluntarily sign the Informed Consent Form prior to participating in any study-specific procedures or assessments
* Depression (PHQ-9 >= 10 and functional impairment present indicated with "difficulty" question OR sufficiently depressed to be enrolled in rTMS therapy)
* Confirmed diagnosis of Major Depressive Disorder (MDD)
* Can maintain all existing treatments (e.g. psychopharmacology, psychotherapy, etc.,) throughout course of the three sessions (psychological / functional assessments, MRI, and TMS), with modifications only as needed for clinical management
* Is a Veteran

Cohort 2:

* Between 18 and 89 years of age
* Ability to safely and comfortably undergo an MRI and tES
* Ability to read, verbalize, understand, and voluntarily sign the Informed Consent Form prior to participating in any study-specific procedures or assessments
* Depression (PHQ-9 >= 10) and endorse that the COVID-19 pandemic has worsened their depression OR have a score on the COVID Stress Scale (CSS) on any item of 3 or greater indicating stressor is "very" or "often" a problem will allow the Veteran to enter the study

Exclusion Criteria:

* Participants who can not safely and comfortably undergo MRI OR TMS (or TES for Cohort 2)
* If their language is not primarily English they may be excluded depending on how dependent the imaging and cognitive tasks are on language

  * Additionally, participants may be excluded if they do not fully understand the consenting process and cannot communicate sufficiently in English to participate in the therapy (d/t language barrier, etc.)
  * An example of safety screen details for an MRI is detailed in the Stanford University MRI screening form
* MRI exclusions include having any non-removable device or implant that makes scanning unsafe, claustrophobia, and size (e.g. weight, girth) beyond the constraints of the MRI and scanner bed
* For TMS the investigators will follow safety guidelines set by Rossi et. al.,2009

  * Specifically, the investigators will not include subjects whose Motor Threshold (MT) is greater than 84% of maximum device output because mathematically they would not be able to be safely stimulated using the standard 120% of MT (i.e. the device cannot stimulate more than 100% of its potential output)
  * The investigators will report these high MT data in our secondary analyses. Additional TMS exclusions include any history or condition that puts patients at risk for a seizure
* Pregnant or planning to become pregnant within the next 3 months
* Lifetime history of moderate or severe traumatic brain injury, current unstable medical conditions, current (or past if appropriate) significant neurological disorder, or lifetime history of:

  * seizure disorder
  * primary or secondary CNS tumors
  * stroke
  * cerebral aneurysm
* Significant cognitive impairment (Montreal Cognitive Assessment [MoCA] < 16)
* Comorbidities (e.g. PTSD) determined not to be the primary diagnosis
* Have a lifetime diagnosis of schizophrenia, schizoaffective disorder, schizophreniform, delusional disorder, or current psychotic symptoms
* Have a diagnosis of obsessive-compulsive disorder assessed by a study investigator to be causing greater impairment than MDD
* Have active suicidal intent or plan in which case Dr. Rosen will determine whether the patient needs to be referred for hospitalization
* Presence of any other condition or circumstance that, in opinion of the investigator team, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments

Exclusion Criteria for Cohort 2:

* Participants who cannot safely and comfortably undergo MRI or TES
* Pregnant or lactating female or planning to become pregnant within the next 3 months
* Lifetime history of moderate or severe traumatic brain injury or tumor
* Significant cognitive impairment (Montreal Cognitive Assessment [MoCA] < 16 OR equivalent score on [MoCA-BLIND] and judgement of a clinician that the test is validly reflecting a significant disabling cognitive impairment
* Have a lifetime diagnosis of:

  * schizophrenia
  * schizoaffective disorder
  * schizophreniform
  * delusional disorder
  * or current psychotic symptoms
* Have a diagnosis of obsessive-compulsive disorder or unstable substance use disorder
* Presence of actively infections/contagious disease such as the flu or SARS-CoV-2

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veteran patients with depression or COVID-19-related distress
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 | Baseline
  Assessment of global functioning. Range from 0 to 100 (0 = no disability, 100 = full disability).
Veterans RAND 36-Item | Baseline
  Assessment of self-reported health-related quality of life. Physical and Mental Component Scores (PCS and MCS) are normed (x = 50, sd = 10) and range from 0 to 100 (0 = worst health, 100 = best health).

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale-17 Items (HAMD-17) | Baseline
  Clinician administered depression symptom assessment scale. Total score ranges from 0 (no depressive symptoms) to 52 (severe depressive symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Allyson C Rosen, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
We are sharing with collaborating institutions.